CLINICAL TRIAL: NCT07331337
Title: Effectiveness of Scapular Strengthening on Pain, Grip Strength, and Function in Chronic Lateral Epicondylitis
Brief Title: Scapular Strengthening Exercises in Patients With Chronic Lateral Epicondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Researcher, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-03/MPT-2020/MSK/CIHS
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Lateral Epicondylitis
Keywords: Conventional Therapy; Scapular Strength; Grip Strength; Functional Ability; Pain; Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow; Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular Strengthening (Experimental): The experimental group received scapular strengthening in addition to conventional therapy.
  Interventions: Other: Scapular strengthening and conventional therapy
- Conventional Therapy (Active Comparator): The control group received conventional therapy.
  Interventions: Other: Conventional Therapy

INTERVENTIONS:
Other: Scapular strengthening and conventional therapy — Scapular strengthening, along with conventional therapy that consisted of ultrasound therapy and static stretching.
  Arms: Scapular Strengthening
Other: Conventional Therapy — Conventional therapy consisted of ultrasound therapy and static stretching.
  Arms: Conventional Therapy

SUMMARY:
Lateral epicondylitis is a prevalent musculoskeletal disorder, affecting 1-3% of the population, typically in middle age and without gender bias. Evidence on the role of scapular strengthening in managing pain, grip strength, and functional limitations in these patients remains limited. This study investigated the impact of scapular muscle strengthening combined with conventional therapy versus conventional therapy alone on these outcomes in individuals with chronic lateral epicondylitis. Thirty participants were randomly assigned to either a control group or an experimental group. Pain was assessed using the visual analogue scale, grip strength with a handheld dynamometer, and functional limitation with the patient-rated tennis elbow (PRTE) scale. The independent variables were the two treatment approaches: conventional therapy alone and conventional therapy supplemented with scapular strengthening.

ELIGIBILITY:
Inclusion Criteria:

* Chronic lateral epicondylitis,
* Positive Mill's test.

Exclusion Criteria:

* Fracture in the shoulder, wrist, or elbow region,
* Upper motor neurological disorder,
* Fibromyalgia,
* Cervical radiculopathy,
* Recent burn,
* Peripheral neuropathy,
* Any surgery on the upper quadrant within six months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-10-23 (Actual)

PRIMARY OUTCOMES:
Pain at elbow | 4 weeks
  Pain will be measured using the Visual Analogue Scale. This scale has a minimum value of 0 and a maximum value of 10. A higher score means a worse outcome.

SECONDARY OUTCOMES:
Grip strength | 4 weeks
  Grip strength will be measured using a Jamar Hydraulic Hand Dynamometer
Functional difficulty | 4 weeks.
  Functional difficulty will be measured using the Patient-Reported Tennis Elbow Evaluation (PRTE) scale. This scale ranges from a minimum of 0 (no pain or disability) to a maximum of 100 (worst pain and disability imaginable). A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th., Principal Investigator — King Saud University
Locations (1):
- Cooperative Institute of Health Sciences, Thalassery, Kannur, Kerala, India

IPD SHARING:
Plan to Share IPD: No